CLINICAL TRIAL: NCT03849248
Title: The Effect of Maternal Scent on Nutrition and Development of Preterm Infants
Brief Title: Maternal Scent and Preterm Infant Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Lama Charafeddine, Associate Professor of Pediatrics and Neonatology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SBS-2018-0527
Record Dates: First submitted 2019-01-24; First posted 2019-02-21 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Behavior, Infant; Development, Infant; Development, Child
Keywords: maternal scent; infant behavior; feeding patterns; stress levels
MeSH Terms: conditions — Infant Behavior; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group of babies will have a maternal scented cloth placed under their heads
  Interventions: Other: Maternal scent cloth
- Control (No Intervention): This group of babies will have a clean non- maternal scented cloth placed under their head

INTERVENTIONS:
Other: Maternal scent cloth — The babies assigned to the intervention group will have a cloth with their mother's scent on it placed under their heads.
  Arms: Intervention

SUMMARY:
To study the effect of maternal scent on the oral feeding, behavior and stress level of premature infants hospitalized in the Neonatal intensive care unit and to assess its potential effect on their development at 18 to 24 months.

DETAILED DESCRIPTION:
Premature infants develop their sense of smell very early in the womb. After birth infants can recognize and distinguish the odor of their mother from their father and others. Premature infants are capable of smelling and they experience less pain and agitation when they smell their mother's milk; studies have shown that premature infants have better sucking and feeding, and they may go home earlier when they are exposed to the odor of breast milk. It is not known whether the same will happen if preterm infants are exposed to their mother's smell rather than the smell of the maternal milk.

ELIGIBILITY:
Inclusion Criteria:

* Mother of a baby who was born premature before completing 36 weeks of pregnancy
* Baby between ages of 5-10 days
* Medically stable baby
* Baby already began feeding by mouth or by feeding tube

Exclusion Criteria:

* Medically unstable baby born after 36 weeks of gestation.

Ages: 5 Days to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2019-05-24 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Salivary cortisol level | Two years
  The saliva will be collected from infant mouth after enrollment the first day before placing the scented cloth under the infant's head and the second after the exposure to the second cloth.
  Levels will be compared before and after and between groups.

SECONDARY OUTCOMES:
Physiological parameters: Heart rate and respiratory rate | Two years
  Infant's heart rate and respiratory rates will be measured.
Achievement of oral feeding | Two years
  The number of days to reach oral feeding of all prescribed feeds will be recorded from the infant medical record, this will be compared between the intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Lama Charafeddine, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon